CLINICAL TRIAL: NCT07213271
Title: The Impact of Dance Intervention on Metabolic Health, Gut Microbiota, Physical Fitness, and Quality of Life in Obese Breast Cancer Survivors
Brief Title: Physical Exercise on Metabolic Health, Gut Microbiota, Physical Fitness, and Quality of Life in Obese Breast Cancer Survivors
Acronym: OBINT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Principal Investigator, Viktor Bielik, professor, Comenius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APVV-22-0047
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Females

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance (Experimental): The patients engaged in dance classes two times a week for 3 months
  Interventions: Other: Dance classes
- Patients without organized physical exercise (No Intervention): The patients engaged in no structured or self-induced physical exercise or activity (sedentary individuals)

INTERVENTIONS:
Other: Dance classes — Participants will attend supervised sessions three times per week, each lasting 60 minutes. Classes were instructed by certified professional dancers and incorporated structured choreographies from three dance genres: folkloric, Latin American, and contemporary.
  Arms: Dance

SUMMARY:
The goal of this clinical trial is to evaluate whether a 3-month dance-based exercise program combined with individualized nutrition can improve health outcomes in obese breast cancer survivors in remission. The main questions it aims to answer are:

Will the intervention reduce body weight, body fat, and visceral adiposity?

Will it improve cardiorespiratory fitness, motor performance, gut microbiota composition, and quality of life?

Researchers will compare women participating in the dance and nutrition program with a control group who maintain their usual lifestyle to see if the intervention leads to favorable metabolic, physical, and microbiome-related changes.

Participants will:

Attend supervised dance classes three times per week for 12 weeks.

Follow an individualized nutrition plan tailored to their resting metabolic rate.

Provide blood and stool samples, complete fitness tests, and answer quality-of-life questionnaires before and after the intervention.

DETAILED DESCRIPTION:
Breast cancer is one of the most prevalent cancers worldwide and its survivors frequently face long-term challenges even after successful treatment. Obesity is a well-established risk factor for both the development and recurrence of breast cancer, and it often worsens treatment-related side effects. Furthermore, increasing evidence suggests that obesity and breast cancer therapies can disrupt the gut microbiota, which may contribute to metabolic complications, systemic inflammation, impaired immunity, and reduced quality of life. Effective, non-pharmacological strategies that simultaneously target metabolic health, microbiome recovery, and physical function are needed for this growing patient population.

The present randomized controlled trial has been designed to examine whether a dance-based physical activity intervention combined with individualized nutrition can favorably influence metabolic health, gut microbiota composition, physical fitness, and quality of life in obese breast cancer survivors in remission. Dance was chosen as the primary exercise modality because it integrates aerobic, strength, and motor-coordination elements in an engaging and culturally adaptable format that may enhance adherence compared to conventional exercise programs.

A total of approximately 40 women with a history of breast cancer, currently in remission and classified as obese, will be recruited and randomized into two groups: an intervention group and a control group. The intervention group will participate in supervised dance sessions three times per week, each lasting 60 minutes, for a total of 12 weeks. Classes will be delivered by certified professional instructors and will include choreographies from folkloric, Latin American, and contemporary dance. To further support metabolic improvements, participants in this group will also receive a personalized dietary plan generated using specialized software, prescribing an energy intake of 1200-1500 kcal/day with balanced proportions of carbohydrates (30-50%), fats (25-30%), proteins (20-30%), and fiber (14 g/1000 kcal). The control group will be instructed to continue their usual daily routines and refrain from initiating new structured physical activities during the study period.

Before and after the intervention, all participants will undergo comprehensive evaluations, including:

* Anthropometry and body composition (weight, BMI, fat mass, visceral fat, waist-hip ratio, muscle mass, resting metabolic rate) using validated bioimpedance and anthropometric methods.
* Physical fitness testing, including a maximal cardiopulmonary exercise test on a cycle ergometer to determine VO₂max, ventilatory parameters, and workload capacity, along with motor performance assessments (handgrip strength, 30-second chair stand, and 30-second arm curl tests).
* Biochemical analysis, including fasting glucose, insulin, lipid profile, liver enzymes, and insulin resistance index (HOMA-IR).
* Gut permeability assessment through serum zonulin measurements.
* Gut microbiota profiling using 16S rRNA sequencing of fecal samples, with alpha and beta diversity indices and taxonomic composition analyses.
* Dietary intake assessed by 3-day food diaries analyzed for caloric and nutrient content.
* Quality of life measured using the EORTC QLQ-C30 and the breast cancer-specific BR23 questionnaire.

The primary outcomes of interest will be changes in body composition (weight, BMI, fat and visceral adiposity) and cardiorespiratory fitness (VO₂max). Secondary outcomes include alterations in gut microbiota diversity and community structure, gut permeability, metabolic biomarkers, dietary patterns, motor performance, and quality-of-life scores. It is hypothesized that obese breast cancer survivors participating in the dance and nutrition program will show:

1. Reductions in body weight, BMI, and fat mass compared to controls.
2. Improvements in cardiorespiratory fitness and muscle endurance.
3. Favorable modifications in gut microbiota composition and diversity.
4. Enhanced quality of life, particularly in physical, emotional, and social domains.

The findings of this study are expected to contribute to a deeper understanding of the role of structured physical activity and diet in post-cancer recovery. Specifically, this trial will provide novel evidence on how a culturally engaging, sustainable, and enjoyable form of exercise - dance - combined with individualized nutrition may promote metabolic health, microbiome restoration, and long-term well-being in obese breast cancer survivors. If effective, this intervention model could be implemented in rehabilitation programs and community health settings to support survivorship care and reduce the risk of cancer recurrence and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer disease
* At least one year after breast cancer treatment
* Must be able to swallow tablets
* Must be able to folow physical exercise training

Exclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Insulin dependent diabetes
* Infectious diseases within the past 2 months
* Use of antibiotics within the past 4 weeks before recruitment

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota Composition (alpha and beta diversity indices) | Baseline to 12 weeks
  Evaluated using 16S rRNA sequencing of fecal samples; primary indices include Shannon diversity, Chao1 richness, and Bray-Curtis dissimilarity
Metabolite outcome measures | Baseline to 12 weeks
  Systemic inflammation and gut-related metabolites will be assessed by measuring blood biomarkers (hs-CRP, IL-6, TNF-α), fecal inflammatory markers (calprotectin, lactoferrin), and microbiota-derived metabolites including short-chain fatty acids (acetate, propionate, butyrate) in feces and plasma, as well as plasma metabolites such as TMAO and selected bile acids. Intestinal permeability will be evaluated through serum zonulin levels. Together, these measures will provide an integrated view of inflammatory status, microbial metabolic activity, and gut barrier function.
Quality of Life assesment | Baseline to 12 weeks
  Change in Quality of Life (EORTC QLQ-C30 Global Health Score) measured using the EORTC QLQ-C30 questionnaire (version 3.0), with scores transformed to a 0-100 scale according to the scoring manual.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness | Baseline to 12 weeks
  Change in Cardiorespiratory Fitness (VO₂max, ml/min/kg) determined by incremental cardiopulmonary exercise testing on a cycle ergometer to evaluate aerobic capacity.
Body composition | Baseline to 12 weeks
  Change in Fat Mass and Visceral Adiposity measured by bioimpedance (InBody 230 device) to assess reduction in total fat mass and visceral fat levels.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Bielik, PhD, Principal Investigator — Comenius University, Faculty of Physical Education and Sport
Locations (1):
- Comenius University in Bratislava, Faculty of physical education and sport, Bratislava, Slovakia